CLINICAL TRIAL: NCT04111237
Title: Rescuer Fatigue Using Two Thumb Versus Two Finger Method During Simulated Neonatal Cardiopulomnary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Principal Investigator, University College Cork
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: ECM 4(ff) 07/03/18
Record Dates: First submitted 2018-06-27; First posted 2019-10-01 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Cardiac Output, High
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Who Masked: Participant
Masking Description: measuremenst of CO are masked from participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two Finger (Active Comparator): two finger method for performing chest compressions
  Interventions: Behavioral: Two Thumb Technique
- Two Thumb Technique (Experimental): Two Thumb Technique
  Interventions: Behavioral: Two Finger technique

INTERVENTIONS:
Behavioral: Two Finger technique — two finger method for chest compression provuision
  Arms: Two Thumb Technique
Behavioral: Two Thumb Technique — Two thumb technique
  Arms: Two Finger

SUMMARY:
The majority of newborns transition successfully from intrauterine to extrauterine life without any assistance. Less than 1% of all newborns will require extensive neonatal resuscitation involving chest compressions (CC) and medications at birth 1. Chest compressions are indicated for those newborns whose heart rate remains less than 60 beats per minute despite adequate ventilation 1. The American Heart Association (AHA) identifies two different methods of delivering chest compressions; a) the two-thumb (TT) method and b) the two-finger (TF) method. The two-thumb method is favoured by the AHA as it results in higher blood pressure and coronary perfusion pressures and can also be delivered from the head of the bed during umbilical catheter insertion 1.

The quality of CC plays a vital role in delivering effective cardiopulmonary resuscitation (CPR). Solevag et al. report that high-quality CC requires (A) optimal compression:ventilation (C:V) ratio, (B) adequate CC rate, (C) depth of CC as well as (D) full recoil between compressions 2. The American Heart Association (AHA) recommend delivering chest compressions on the lower third of the sternum to a depth of one third the anterior-posterior (AP) chest diameter. The recommended C:V ratio is 3:1 (90 compressions and 30 breaths per minute) 1.

A number of studies have highlighted the effects of rescuer fatigue on quality of chest compressions. One study reported adverse effects on CC quality when performed without interruption over a 3 minute period 6. It has therefore been recommended to rotate rescuers every 2-3 minutes in order to avoid rescuer fatigue and to ensure high quality CC6-7. As well as duration of CC, other factors can contribute to greater levels of rescuer fatigue. A number of studies have looked at the effect of different CC to ventilation methods on rescuer fatigue. Bodingh et al investigated this during simulated infant CPR. They reported greater levels of rescuer fatigue during simulated CPR in CCaV (continuous CC with asynchronous ventilation) at 120 CC per min compared to the recommended 3:1 C:V CPR 3. A similar study was performed by Li et al where rescuer fatigue was assessed during (i) 3:1 C:V ratio, (ii) CCaV at 90 CC per min and (iii) CCaV at 120 CC per min. However, unlike Bodingh et al, they found both 3:1 C:V and CCaV CPR to be equally fatiguing 4. Different CC techniques (TT vs TF method) can also cause varying levels of rescuer fatigue. In a recent study, Jiang et al compared the TT and TF chest compression techniques on infant mannequins and found that the TF method caused greater levels of rescuer fatigue compared with the TT method 5. We therefore set out to investigate whether different CC techniques cause different levels of rescuer fatigue during neonatal CPR. We hypothesize that performing TF method on neonatal mannequins will produce greater levels of rescuer fatigue. The results of this study would have significant implications in terms of choice of CC technique in new-born resuscitation.

The purpose of this study is to compare rescuer fatigue during simulated neonatal chest compressions using two different CC methods; the two-finger (TF) method vs two-thumb (TT) method. This will be performed on both preterm and term mannequins by neonatologists and level of fatigue will be assessed by measuring change in cardiac output during chest compressions.

Hypothesis: Performing CC using the two-finger (TF) method produces higher levels of rescuer fatigue compared with the two-thumb (TT) method during 5 minutes of simulated neonatal CPR.

DETAILED DESCRIPTION:
Inclusion criteria

1. Neonatology NCHD's from CUMH
2. Participants must have completed Neonatal Resuscitation Programme (NRP)
3. Participants must be working as doctors in the area of neonatology Exclusion criteria

1. Any history of cardiac or respiratory disorder 2. Physicians who are post-call/sleep deprived

Intervention:

This will be a crossover trial. Each participant will be assigned to performing ether TT or TF chest compressions. The participant will each perform 5 minutes of simulated chest compressions either a term or preterm mannequin using 3:1 C:V CPR. Each participant will have NICOM leads attached to their body which will record HR and cardiac output. One week later the participant will cross over and perform the alternate CC technique. The trial will initially be performed on a term mannequin for the first 2 weeks before being repeated on a preterm mannequin.

Data Collection:

Recorded data will include: Age, gender, ethnicity, weight, height, BMI, HR and cardiac output. Participants will have an allocated study number, ensuring that the data collected will be anonymised. The list of study numbers and data will be stored in a secure password protected database in the Neonatal Unit. Only people involved in the study and other authorised persons will have access to this information.

Outcome Measures:

Primary Outcome Measure:

Percentage change in cardiac output after 5 minutes of simulated neonatal CPR using two different chest compression methods (2-finger method vs. 2-thumb method) on term and preterm mannequins.

Secondary Outcome Measure:

Perceived level of fatique. At the end of the study session each subject will complete a Likert scale-based questionnaire on subjective feeling of fatigue.

ELIGIBILITY:
Inclusion Criteria:

Neonatology NCHD's from CUMH

Participants must have completed Neonatal Resuscitation Programme (NRP)

Participants must be working as doctors in the area of neonatology

Exclusion Criteria:

Any history of cardiac or respiratory disorder

Physicians who are post-call/sleep deprived

Pregannt

Ages: 24 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage change in cardiac output after 5 minutes of simulated neonatal CPR | 1 month
  using two different chest compression methods (2-finger method vs. 2-thumb method) on term and preterm mannequins.

CONTACTS AND LOCATIONS:
Locations (1):
- UCC, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No